CLINICAL TRIAL: NCT03994614
Title: The Clinical Trial of the Effect of Transcutaneous Electrical Acupoint Stimulation on the Quality of the Oocyte on Poor Ovarian Response
Brief Title: the Effect of Transcutaneous Electrical Acupoint Stimulation on the Quality of Oocyte on Poor Ovarian Response(POR)
Acronym: POR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ShangHai Ji Ai Genetics & IVF Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JIAI 2019-4
Record Dates: First submitted 2019-04-02; First posted 2019-06-21 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Poor Ovarian Response
Keywords: transcutaneous electrical acupoint stimulation; quality of oocyte; ovarian reserve; poor ovarian response; in vitro fertilization-embryo transfer

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the TEAS intervention group (Experimental): Patients in this group will be given TEAS treatment for 12 weeks prior to COS.
  Interventions: Other: TEAS
- No intervention group (No Intervention): Patients in this group will not be given any interventions for 12 weeks prior to COS.

INTERVENTIONS:
Other: TEAS — Patients in the experimental group will be given TEAS treatment for 12 weeks prior to COS. The patients will be given three times acupuncture every week except menstruation. The acupuncture acupoint locations are as follows: head acupoint Baihui(DU20), abdominal acupoint Zhongji (RN3), Guanyuan (RN4), Zigong(EX-CA1), leg acupoint Sanyinjiao(SP6), waist acupoint Shenyu (BL23) and Guanyuanyu(BL26).
  Arms: the TEAS intervention group

SUMMARY:
Patients in experimental group will be given transcutaneous electrical acupoint stimulation (TEAS) treatment for 12 weeks prior to controlled ovarian stimulation (COS).The patients will be given three times acupuncture every week except menstruation.Patients in no intervention group will not be given any interventions for 12 weeks prior to COS. The primary outcome measure is the number of MII eggs obtained in the COS cycle. The secondary outcome measures are the lab and clinical reproductive outcomes.

DETAILED DESCRIPTION:
The patients will be randomly recruited into two groups. Patients in experimental group will be given TEAS treatment for 12 weeks prior to COS.The patients will be given three times acupuncture every week except menstruation. One treatment lasts for 30 minutes. The acupoints used for the TEAS treatment included head acupoint Baihui(DU20), abdominal acupoint Zhongji (RN3), Guanyuan (RN4), Zigong(EX-CA1), leg acupoint Sanyinjiao(SP6), waist acupoint Shenyu (BL23) and Guanyuanyu(BL26). Patients in no intervention group will not be given any intervention for 12 weeks prior to COS. When at least one dominant follicle is greater than 18 mm then injection a GnRH agonist (Triptorelin, Ferring, Switzerland) 0.2mg. 36 hours later transvaginal oocyte retrieval will be taken. After 3 hours of incubation, each egg will be transferred with a density of about 100,000/mllive sperm. The fresh embryo transfer is performed 72 hours after embryo culture in vitro. The whole embryos will be frozen.

The primary outcome measure is the number of MII eggs obtained in the COS cycle. The secondary outcome measures are the lab and clinical reproductive outcomes,including basic endocrine, serum Anti-Mullerian Hormone （AMH）, antral follicle counts, fertilization rate, cleavage rate, number of D3 embryos, the clinical pregnancy rate and early abortion rate.

ELIGIBILITY:
Inclusion Criteria:

1. The poor ovarian response patients compliance with Bologna consensus
2. Age：20-45 year
3. Women undergoing IVF-ET because of infertility for more than one year.

Exclusion Criteria:

1. Patients with genital tract malformation. Uterine malformation (single uterus, double uterus, double uterus, untreated mediastinal uterus) and other effects affecting uterine cavity disease (adenomyosis, submucosal uterine fibroids, intrauterine adhesions and scar uterus)
2. Complicated with other medical diseases（Hypertension, diabetes, psychosis, hereditary diseases）

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 92 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
The number of MII eggs | one day after oocyte pickup
  The number of MII eggs obtained in the COS cycle

SECONDARY OUTCOMES:
Basic Follicle stimulating hormone （FSH） value | On Day two of menstruation
  Basic FSH value in mIU/ml
Basic Luteinizing hormone （LH） value | On Day two of menstruation
  Basic LH in mIU/ml
Basic estrodiol value | On Day two of menstruation
  Basic estrodiol in pg/ml
Serum AMH value | On Day two of menstruation
  Serum AMH in ng/ml
antral follicle count | antral follicle count On Day two of menstruation
  antral follicle count
fertilization rate | fertilization rate calculated on 1 day after oocyte pickup
  fertilization rate
cleavage rate | cleavage rate calculated on 2 days after oocyte pickup
  cleavage rate
the number of Day 3 embryos | the number of Day 3 embryos calculated on 3 days after oocyte pickup
  the number of Day 3 embryos
clinical pregnancy rate | clinical pregnancy rate calculated on the 6th gestational week
  clinical pregnancy rate
early abortion rate | early abortion rate calculated on 12th week of pregnancy
  early abortion rate

CONTACTS AND LOCATIONS:
Overall Officials: Wenbi Zhang, doctor, Principal Investigator — Fudan University
Locations (1):
- Shanghai Ji Ai Genetics & IVF Institute, Obstetrics and Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No